CLINICAL TRIAL: NCT04273568
Title: The Effect of Scapular Proprioceptive Neuromuscular Facilitation Techniques on Pain and Functionality in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Akgüller (Other)
Responsible Party: Sponsor-Investigator, Tuğba Akgüller, Lecturer, Istanbul Arel University
Organization: Istanbul Arel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tugbaakguller
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Proprioceptive Neuromuscular Facilitation; Shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (PNF group) (Experimental): Scapular PNF and exercise program was applied to the PNF group.
  Interventions: Other: Scapular PNF; Other: Exercise program
- Group 2 (Exercise group) (Active Comparator): Exercise program was applied to the exercise group
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Scapular PNF — Rhythmic initiation and repetitive stretching techniques in scapula anterior elevation-posterior depression and anterior depression-posterior elevation patterns were applied twice a week for 6 weeks.
  Arms: Group1 (PNF group)
Other: Exercise program — An exercise program consisting of exercises used in the conservative treatment of shoulder impingement syndrome for both groups was applied twice a week for 6 weeks.

SUMMARY:
The aim of this study was to investigate the effects of scapular proprioceptive neuromuscular facilitation (PNF) techniques applied in addition to exercise therapy in patients with Subacromial impingement syndrome (SIS) on pain, pressure pain threshold (PPT), range of motion (ROM), functionality, scapular dyskinesis, active trigger points and emotional state.

DETAILED DESCRIPTION:
32 patients between the ages of 20-60 diagnosed with SIS were included in the study.

The patients were randomly divided into two groups. The exercise group received an exercise program of 12 sessions. Scapular PNF techniques were applied to the PNF group with the same exercise program. Patients were evaluated twice; one before and one after 6 weeks of treatment; using Visual Analogue Scale (VAS) for pain, algometer for PPT, digital goniometer for range of motion (ROM), The Disabilities of Arm, Shoulder and Hand (DASH) for functional status, lateral scapular slide test (LSST) for scapular dyskinesis, Travell and Simons criteria for trigger point and Hospital Anxiety and Depression Scale (HADS) for emotional state. At the end of treatment patient satisfaction was evaluated with Global Change Scale.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 60
* Diagnosed with SIS by MRI and clinical examination and a specialist physician
* Positive impingement tests (Hawkings, Neer and Jobe test) or painful motion arc (60 ° -120 °)
* Unilateral shoulder pain that has been going on for at least 3 months
* Signed voluntary consent form

Exclusion Criteria:

* Diagnosed with adhesive capsulitis or massive rotator cuff tear
* Having undergone upper limb surgery
* Presence of rheumatological systemic diseases
* Presence of Glenohumeral instability
* Having a neurological disease affecting the upper extremity
* Diagnosed with cervical radiculopathy
* Degenerative joint disorders
* Having communication problems
* Steroid injection therapy or physiotherapy in the past 6 months have been rehabilitated

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain intensity of the patients at 6 weeks | Baseline and 6 weeks
  Pain intensity of the patients at rest, during activity and at night was assessed using the VAS; Visual Analog Scale. In this evaluation, individuals were told that the number "0" on the 10 cm long horizontal line expresses "no pain", and the number "10" indicates "unbearable pain" and that individuals should mark their intensity of pain on this line.
Change from Baseline Functional Status of the patients at 6 weeks | Baseline and 6 weeks
  The functional status of the patients were evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH). DASH is a scale consisting of 30 questions that question the functional status and symptoms used in musculoskeletal disorders of the upper extremity.The number of Likert scale (1: no difficulty, 5: I can not do at all) is used in answering the questions and the total score obtained is between 0 and 100.

SECONDARY OUTCOMES:
Shoulder Range of Motion (ROM) | Baseline and 6 weeks
  EHA evaluations of flexion, abduction, internal rotation and external rotation of the shoulder joint were performed in the supine position using the digital goniometer.
Pain Pressure Threshold (PPT) | Baseline and 6 weeks
  Pressure pain threshold was evaluated using the Algometer (dolorimeter).
Scapular dyskinesis | Baseline and 6 weeks
  Scapular Dyskinesis was evaluated with "The Lateral Scapular Slide Test (LSKT)". In this test, the distance of the inferior angle of the scapula to the nearest spinous process at 3 different positions (0°, 40-45°, 90°) is measured, and a difference of 1 cm or more between the two sides in any of the three positions is considered positive for scapular dyskinesis.
Active trigger points | Baseline and 6 weeks
  Active trigger points were evaluated by palpation method according to Travell and Simons criteria. Scalene, upper trapezius, levator scapula, supraspinatus, infraspinatus, subskapularis, teres minor, teres major, deltoid anterior, middle and posterior group fibers, pectoralis major, pectoralis minor, biceps brachii muscles were evaluated with palpation method in terms of trigger point presence.
Emotional state | Baseline and 6 weeks
  The emotional states of the cases were evaluated using the Hospital Anxiety and Depression Scale (HAD), which consists of 14 questions. (HAD). This scale has a 7-question anxiety (HAD-A) subscale that evaluates the anxiety state, and a 7-question depression (HAD-D) subscale that evaluates the state of depression, and a four-point likert scale is used to answer the questions. For the total score of each sub-score, 0-7 points are normal, 8-10 points are at the border, and 11 points are defined as abnormal

OTHER OUTCOMES:
Patient Satisfaction: Global Rating of Change (GRC) scale | At the end of the 6-weeks treatment
  Patient Satisfaction was assessed Global Rating of Change (GRC) scale. The scale used included 5 points (-2: I am much worse. -1: I am worse, 0: I am the same, +1: I am better, +2: I am much better).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)